CLINICAL TRIAL: NCT03884192
Title: CONSIST: A Phase III Randomized Control Study of Consolidation Sintilimab (IBI308) After Concurrent Chemoradiation Versus Chemoradiation Alone in Patients With Unresectable Local Advanced Stage III NSCLC
Brief Title: Consolidation Sintilimab After Concurrent Chemoradiation in Patients With Unresectable Stage III NSCLC
Acronym: CONSIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONSIST
Record Dates: First submitted 2019-01-11; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Locally advanced; Stage III Non-Small Cell Lung Cancer; Unresectable Non-Small Cell Lung Cancer; Concurrent Chemoradiation; Immune-mediated cancer therapy; PD-1; Sintilimab; IBI308
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab Arm (Experimental): Sintilimab consolidation therapy
  Interventions: Drug: Consolidation Sintilimab
- Observation Arm (No Intervention): Observation

INTERVENTIONS:
Drug: Consolidation Sintilimab — Sintilimab consolidation therapy after concurrent chemoradiation, 200mg IV, every 3 weeks, until progressive disease (PD, unless patients can continuously benefit from study treatment per investigators' judgement), start new anti-cancer therapy, intolerable toxicity, withdraw informed consent or other conditions that require study treatment discontinuation. Sintilimab will be given at a maximum of 12 months.
  Arms: Sintilimab Arm

SUMMARY:
This is an open label, multi-center, randomized, control phase III trial, to compare the efficacy and safety of consolidation therapy with sintilimab (IBI308) versus best supported care (BSC), in unresectable stage III NSCLC patients who do not experience disease progression after initial concurrent chemoradiation.

DETAILED DESCRIPTION:
This is an open label, multi-center, randomized, control study of sintilimab versus BSC in unresectable local advanced stage III NSCLC patients without disease progression after concurrent chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before initiation of any study procedures
2. Age ≥ 18 years and ≤ 75 years
3. Histologically or cytologically confirmed NSCLC, with unresectable local advanced disease (stage III according to NSCLC staging version 8)
4. Expected survival over 3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
6. At least 1 measurable disease according to RECIST 1.1
7. Pulmonary function: forced expiratory volume at one second (FEV1) > 1 liter(L)
8. Patient must not have received any anti-cancer therapy for the purpose of treating lung cancer. However, exploratory thoracotomy, mediastinoscopy, excision biopsy, and other kinds of surgery for diagnosis and staging purpose is acceptable. Patients with local or regional recurrent disease after pneumonectomy is allowed to participate if they meet other inclusion criteria (e.g. stage III, inappropriate for re-operation).
9. For all female patients of childbearing potential, a negative pregnancy test (either urine or serum) must be obtained within 3 days before the first dose (Cycle 1, Day 1) of study treatment. If a urine pregnancy test shows an unconfirmed result, a serum pregnancy test must be performed.
10. Adequate hematopoietic function, defined as: absolute neutrophil count (ANC) ≥ 1.5 x 10*9/L; platelet count ≥100 x 10*9/L; hemoglobin ≥90 g/L [no blood transfusion within 7 days or not erythropoietin (EPO) dependent]
11. Adequate liver function, defined as: total serum bilirubin ≤ 1.5 x upper limit of normal (ULN); serum alanine transaminase (ALT) and aspartic transaminase (AST) ≤ 2.5 x ULN, with no liver transplantation
12. Adequate renal function, defined as: serum creatinine ≤ 1.5 x ULN or calculated creatinine-clearance ≥ 60 ml/min (Cockcroft-Gault). Urine protein less than 2+ by urinalysis or 24-hour urinary protein quantity < 1g
13. Adequate coagulation function, defined as: international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN. For patients receiving anticoagulant therapy can be enrolled if PT is within the range defined by anticoagulant therapy.
14. Myocardial enzymes are within normal range
15. All subjects of childbearing potential must agree to use efficient contraceptive methods that result in a failure rate of < 1% per year during the study treatment period and for at least 180 days after discontinuation from study treatment.

Exclusion Criteria:

1. Being treated by other investigational drugs within an interventional study, or have received any investigational drugs or instruments within 4 weeks prior to the first dose of study treatment
2. Being enrolled in other interventional studies, unless they are observational studies or during the follow-up stage of an interventional study
3. NSCLC histology with small cell lung cancer (SCLC) components
4. Active or autoimmune disease history (within the past 2 years), or history of immune deficiency
5. Previous immune therapy including: anti PD-1, anti PD-L1, anti PD-L2 or treatment targeting other co-stimulatory or co-inhibitory T-cell receptors [e.g. cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, and CD137]

   a) Systemic therapy with Chinese patent medicine or drugs of immunoregulation effect (including thymosin, interferon, interleukin, unless local delivery for controlling pleural effusion) within 2 weeks prior to the first dose of study treatment, or major surgery within 4 weeks prior to the first dose of study treatment
6. Clinical evidence of active diverticulitis, abdominal abscess, or gastrointestinal obstruction
7. Previous organ or blood system transplantation
8. Known allergic to pemetrexed, paclitaxel, etoposide, cisplatin, carboplatin, sintilimab component and/or any excipients
9. A history of active autoimmune disease requiring systemic treatment (e.g. using drugs for disease remission, corticosteroids or immunosuppressor) within 2 years prior to the first dose of study treatment. Substitution therapy (e.g. thyroxine, insulin or physiological corticosteroids for treating adrenal or pituitary dysfunction) is not considered as a systemic treatment.

   a) Diagnosis as immunodeficiency, or being treated with systemic glucocorticoid or other kinds of immunosuppressor within 7 days prior to the first dose of study treatment. A physiological dose of glucocorticoid (≤10 mg/day prednisone or equivalent dose of other steroids) is permitted.
10. Previously diagnosis as other malignant tumors within 5 years prior to the first dose of study treatment, with the exception of: skin basal cell carcinoma or squamous cell carcinoma with radical treatment, and/or carcinoma in situ underwent radical resection
11. History of non-infectious pneumonitis requiring treatment with glucocorticoid within 1 year prior to the first dose of study treatment, or currently existed interstitial lung disease
12. Active infectious that required systemic therapy
13. Know psychiatric illness or drug abuse that would limit compliance with study requirements
14. Know human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive)
15. Untreated active viral hepatitis B (HBV)

    Patients with HBV who meet the following criteria are also eligible:
    1. HBV virus load (VL) <1000 copy/ml (200 IU/ml), and patients must continuously receive anti-HBV therapy during all through study treatment phase to prevent virus activation
    2. Patients with a result of anti-HBc(+)、HBsAg (-)、anti-HBs (-) 和 HBV VL (-) are not required to receive prophylactic anti-HBV therapy, but must be closely monitored for virus re-activation
16. Patients with active HCV infection (HCV antibody positive and HCV-RNA > the lower detection limit)
17. History or evidence of disease, treatment or laboratory abnormalities that would interfere the study outcome, prevent patients from participating entirely, or ineligible to enroll per the investigators' judgement
18. Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months after enrollment or study close
  PFS (per RECIST 1.1 as assessed by the investigator) will be defined as the time from the date of randomisation until the date of objective disease progression or death (by any cause in the absence of progression).

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months after enrollment or study close
  OS (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date of randomisation until death due to any cause.
Objective Response Rate (ORR) | up to 24 months after enrollment or study close
  ORR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | up to 24 months after enrollment or study close
  DCR (per RECIST 1.1 as assessed by the investigator) is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR), or stable disease (SD).
Duration of Response (DoR) | up to 24 months after enrollment or study close
  DoR (per RECIST 1.1 as assessed by the investigator) is defined as the time from the date for first documented response of complete response (CR) or partial response (PR) until the date for the first documented response of progressive disease (PD) or death in the absence of progression.
Progression Free Survival (PFS) Rate at 12/18 months | From the date of randomization until the Kaplan-Meier estimate of PFS at 12/18months
  PFS rate at 12/18 months is defined as the proportion (%) of patients who are alive and progression free at 12 and 18months from the date of randomisation.
Treatment-related Adverse Events (AEs) | From the date of randomization to 90 days after last dose of study treatment
  The grade of AEs and the number of patients with AEs are assessed by the investigator based on CTCAE v4.03 from the date of randomization to 90 days after last dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auperin A, Le Pechoux C, Rolland E, Curran WJ, Furuse K, Fournel P, Belderbos J, Clamon G, Ulutin HC, Paulus R, Yamanaka T, Bozonnat MC, Uitterhoeve A, Wang X, Stewart L, Arriagada R, Burdett S, Pignon JP. Meta-analysis of concomitant versus sequential radiochemotherapy in locally advanced non-small-cell lung cancer. J Clin Oncol. 2010 May 1;28(13):2181-90. doi: 10.1200/JCO.2009.26.2543. Epub 2010 Mar 29. PMID 20351327
- [Background] Yoon SM, Shaikh T, Hallman M. Therapeutic management options for stage III non-small cell lung cancer. World J Clin Oncol. 2017 Feb 10;8(1):1-20. doi: 10.5306/wjco.v8.i1.1. PMID 28246582
- [Background] Ahn JS, Ahn YC, Kim JH, Lee CG, Cho EK, Lee KC, Chen M, Kim DW, Kim HK, Min YJ, Kang JH, Choi JH, Kim SW, Zhu G, Wu YL, Kim SR, Lee KH, Song HS, Choi YL, Sun JM, Jung SH, Ahn MJ, Park K. Multinational Randomized Phase III Trial With or Without Consolidation Chemotherapy Using Docetaxel and Cisplatin After Concurrent Chemoradiation in Inoperable Stage III Non-Small-Cell Lung Cancer: KCSG-LU05-04. J Clin Oncol. 2015 Aug 20;33(24):2660-6. doi: 10.1200/JCO.2014.60.0130. Epub 2015 Jul 6. PMID 26150444
- [Background] Ettinger DS, Wood DE, Aisner DL, Akerley W, Bauman J, Chirieac LR, D'Amico TA, DeCamp MM, Dilling TJ, Dobelbower M, Doebele RC, Govindan R, Gubens MA, Hennon M, Horn L, Komaki R, Lackner RP, Lanuti M, Leal TA, Leisch LJ, Lilenbaum R, Lin J, Loo BW Jr, Martins R, Otterson GA, Reckamp K, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer K, Yang SC, Gregory K, Hughes M. Non-Small Cell Lung Cancer, Version 5.2017, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2017 Apr;15(4):504-535. doi: 10.6004/jnccn.2017.0050. PMID 28404761
- [Background] Bradley JD, Paulus R, Komaki R, Masters G, Blumenschein G, Schild S, Bogart J, Hu C, Forster K, Magliocco A, Kavadi V, Garces YI, Narayan S, Iyengar P, Robinson C, Wynn RB, Koprowski C, Meng J, Beitler J, Gaur R, Curran W Jr, Choy H. Standard-dose versus high-dose conformal radiotherapy with concurrent and consolidation carboplatin plus paclitaxel with or without cetuximab for patients with stage IIIA or IIIB non-small-cell lung cancer (RTOG 0617): a randomised, two-by-two factorial phase 3 study. Lancet Oncol. 2015 Feb;16(2):187-99. doi: 10.1016/S1470-2045(14)71207-0. Epub 2015 Jan 16. PMID 25601342
- [Background] Tsujino K, Kurata T, Yamamoto S, Kawaguchi T, Kubo A, Isa S, Hasegawa Y, Ou SH, Takada M, Ando M. Is consolidation chemotherapy after concurrent chemo-radiotherapy beneficial for patients with locally advanced non-small-cell lung cancer? A pooled analysis of the literature. J Thorac Oncol. 2013 Sep;8(9):1181-9. doi: 10.1097/JTO.0b013e3182988348. PMID 23883782
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881